CLINICAL TRIAL: NCT00854893
Title: Enhance of Language Learning with Neurostimulation (transcranial Direct Current Stimulation)
Brief Title: Enhance of Language Learning with Neurostimulation
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Universitätsklinikum Hamburg-Eppendorf (Other)
Collaborators: German Research Foundation (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Crossover | Masking: Triple | Purpose: Treatment
Other Study IDs: PV3128; LI 1892/1-1 (Other Grant/Funding Number: Deutsche Forschungsgemeinschaft (DFG))
Record Dates: First submitted 2009-03-02; First posted 2009-03-03 (Estimated); Last update posted 2024-12-11 (Actual); Status verified 2022-08

CONDITIONS: Stroke; Aphasia; Aging
Keywords: stroke; aphasia; aging; language learning
MeSH Terms: conditions — Stroke; Aphasia | interventions — Transcranial Direct Current Stimulation

STUDY DESIGN:
Who Masked: Participant, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes

ARMS (3):
- anodal (Experimental): anodal stimulation: 20 min during language learning, intensity: 1 mV, anodal electrode over primary motor cortex of language-dominant hemisphere, reference electrode over contralateral supraorbital area
  Interventions: Device: transcranial direct current stimulation
- cathodal (Experimental): anodal stimulation: 20 min during language learning, intensity: 1 mV, cathodal electrode over primary motor cortex of language-dominant hemisphere, reference electrode over contralateral supraorbital area
  Interventions: Device: transcranial direct current stimulation
- sham (placebo) (Experimental): sham stimulation (placebo condition): 30 seconds during language learning, intensity: 1 mV, anodal electrode over primary motor cortex of language-dominant hemisphere, reference electrode over contralateral supraorbital area
  Interventions: Device: transcranial direct current stimulation

INTERVENTIONS:
Device: transcranial direct current stimulation — 1 mV for 20 min (verum conditions: anodal and cathodal)or 30 seconds (placebo condition: sham) during language learning , active electrode over primary motor cortex of language dominant hemisphere, reference electrode over contralateral supraorbital area
  Other Names: DC Stimulator; Manufacturer:eldith -Electro-Diagnostic & Therapeutic Systems GmbH, Gustav-Kirchhoff-Straße 5, D-98693 Ilmenau; Serial number: 0006

SUMMARY:
The purpose of this study is to test the effect of transcranial direct current stimulation over the motor cortex of the language dominant hemisphere on language learning in healthy subjects and stroke patients with aphasia. We hypothesize that anodal stimulation enhances the learning of action words compared to sham and cathodal stimulation.

DETAILED DESCRIPTION:
The motor cortex is involved at different levels of language processing. It has been demonstrated that the perception of action words activates motor representations in the language-dominant hemisphere. However, it is not known whether modulation of excitability has an effect on learning new action words. Thus, we hypothesize that transcranial direct current stimulation over the motor cortex of the language-dominant hemiphere modulates the acquisition of new action words. The results bear the potential to design new rehabilitative strategies in stroke patients with aphasia. The motor cortex might offer an access to the language network that can be used for interventional approaches such as neurostimulation.

ELIGIBILITY:
Inclusion Criteria:

* age >18 and < 86 years
* contractual capability
* ischemic stroke excluding motor cortex (stroke patients)
* minimum time since stroke 9 months
* aphasia (stroke patients)
* severe aphasia that impedes understanding of instructions (stroke patients)

Exclusion Criteria:

* sever head trauma in the past
* seizures
* pace maker
* metal implants in the head/neck region
* severe comorbidity, especially neurologic and psychiatric diseases
* intake of illegal drugs
* Mini Mental State examination score < 27
* neuroactive substances, e.g. antidepressants
* pregnancy

Ages: 18 Years to 86 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 70 (Actual)
Dates: Start 2009-10 (Actual); Primary Completion 2010-01-01 (Actual); Study Completion 2010-07-01 (Actual)

PRIMARY OUTCOMES:
word learning | immediately after intervention and after 1 week
  learning of new action words measured as learned words/all words in %

CONTACTS AND LOCATIONS:
Overall Officials: Gianpiero Liuzzi, MD, Principal Investigator — Universitätskrankenhaus Hamburg-Eppendorf
Locations (1):
- University Hospital Hamburg-Eppendorf, Department of Neurology, Hamburg, Hamburg, Germany

REFERENCES:
- [Background] Branscheidt M, Hoppe J, Freundlieb N, Zwitserlood P, Liuzzi G. tDCS Over the Motor Cortex Shows Differential Effects on Action and Object Words in Associative Word Learning in Healthy Aging. Front Aging Neurosci. 2017 May 15;9:137. doi: 10.3389/fnagi.2017.00137. eCollection 2017. PMID 28555104